CLINICAL TRIAL: NCT06568965
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Arm Clinical Trial of De-Stress and Happy Gut Powder in Relieving Stress and Functional Dyspepsia Symptoms in Adults.
Brief Title: Clinical Study of De-Stress & Happy Gut Powder for Stress and Indigestion in Adults.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herbolab India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHC/CT/24-25/015; CTRI/2024/07/071248 (Registry Identifier: clinical trials registry of India)
Record Dates: First submitted 2024-08-10; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Stress; Dyspepsia; Indigestion
Keywords: stress; Dyspepsia; Indigestion
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Intervention Model Description: Randomized, Double blind, Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- De-stress & happy gut powder-U001 (Experimental)
  Interventions: Other: De-stress & happy gut powder-U001
- De-Stress & Happy Gut powder-I001 (Experimental)
  Interventions: Other: De-Stress & Happy Gut powder-I001
- Placebo Powder 001 (Other)
  Interventions: Other: Placebo Powder 001

INTERVENTIONS:
Other: De-stress & happy gut powder-U001 — Take one sachet daily, 30 minutes before breakfast, for 60 days
  Arms: De-stress & happy gut powder-U001
Other: De-Stress & Happy Gut powder-I001 — Take one sachet daily, 30 minutes before breakfast, for 60 days
  Arms: De-Stress & Happy Gut powder-I001
Other: Placebo Powder 001 — Take one sachet daily, 30 minutes before breakfast, for 60 days
  Arms: Placebo Powder 001

SUMMARY:
The current study focuses on clinical validation of efficacy of nutraceutical product in relieving stress and functional dyspepsia symptoms in adults for gut health. The effect of these nutraceuticals not only targets the physical symptoms but also enhances overall well-being. Improved digestive health leads to better nutrient absorption, which is essential for energy levels and immune function. Reduced stress levels contribute to better sleep quality, cognitive function, and emotional stability.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-arm, clinical trial of De-Stress & Happy Gut powder in relieving stress and functional dyspepsia symptoms in adults.

In this study, more than 81 participants will be enrolled in a 1:1:1 ratio into three groups: Group A (De-stress & Happy Gut Powder-U001), Group B (De-stress & Happy Gut Powder-I001), and Group C (Placebo Powder 001). Each participant will take one sachet daily, 30 minutes before breakfast, for 60 days. The efficacy of the investigational products will be compared between the groups.

Concomitant diseases/medication assessment will be performed on screening. The efficacy of the intervention will be assessed by evaluating changes in the Perceived Stress Scale (PSS) score, Nepean Dyspepsia Index (NDI), changes in serum cortisol levels, changes in the COPE Questionnaire (a. Positive Subscale, b. Denial Subscale) score, assessing gut health using a Gastrointestinal Symptom Rating Scale (GSRS) score will be assessed at screening, day 30, and day 60.

Changes in the State-Trait Anxiety Inventory (STAI) score, changes in the Profile of Mood State (POMS) questionnaire score (a. Total Mood Disturbance, b. Depression) will be assessed at screening and day 60.

Changes in symptom score on a 7-point Likert scale to grade overall symptoms of dyspepsia (Upper abdominal fullness, Pain, Belching, Bloating, Early satiety, Nausea, Vomiting, Regurgitation, Heartburn, Loss of appetite, cravings for junk food) will be assessed at screening, day 15, 30, and day 60.

Changes in gut microbiota at screening and day 60; and time in seconds for relief from pain and heartburn in 5-10 subjects recommended to be used on a need basis in case of acid reflux flare/heartburn will be assessed at baseline, day 15, 30, and day 60.

Treatment compliance, tolerability of investigational products will be assessed at day 30 and day 60. Safety of the investigational treatment in terms of adverse events (AEs), and serious adverse events (SAEs), will be assessed at baseline, day 15, day 30, and day 60.

Assessment of changes in vital sign parameters will be done from screening to end of the study (Day 60).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 21-50 years both inclusive
2. Suffering from self-reported mild to moderate stress on the PSS scale score less than or equal to 26
3. Participants willing to participate in clinical trials and who have read understood and signed the informed consent form
4. No severe anxiety and depression i.e. Generalized anxiety disorder GAD score less than or equal to 10 and Patients' health questionnaire-9 PHQ-9 score less than or equal to 14
5. Diagnosis of functional dyspepsia/non-ulcer dyspepsia by fulfilling Rome-III criteria
6. Participant should be suffering with at least 4 or more symptoms mentioned below and with a total symptom score of 20 or more based on a 7-point Likert scale (a) Upper abdominal fullness (b) Upper abdominal pain (c) Belching (d) Bloating (e) Early satiety (f) Nausea (g) Vomiting (h) Regurgitation (i) Heartburn (j) Loss of appetite

Exclusion Criteria:

1. Inability to perform any of the assessments required for endpoint analysis
2. Known hypersensitivity to investigational products
3. Participants with a history of substance abuse, drugs, heavy use of alcohol, and/or smoking within last 5 years
4. Advanced chronic illness that would impair follow-up or monitoring
5. Participants who have used dietary supplements, medications, such as oral/IV antibiotics or probiotics, or supplements known to affect hunger, satiety, appetite, or gut microbiome within three months prior to recruitment. Additionally, individuals currently using nutraceuticals, allopathic, or ayurvedic supplements for stress and or gastrointestinal health management;
6. Participants suffering from abdominal obesity that is waist circumference of more than 80 cm in females and of more than 90 cm in male;
7. Pregnant or lactating women, as well as women of childbearing potential who are not using contraception or intending to conceive during the study
8. Participants with current or past diagnoses of peptic ulcer disease, gastroesophageal reflux disorder (GERD), or irritable bowel syndrome (IBS), as well as those who have undergone surgery related to these conditions
9. Have any other neurodegenerative diseases, mental illness or dementia
10. Any other clinical condition in the judgment of investigator finds the study participation unsuitable for the participant.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Screening, day 30 and day 60
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress. PSS-10 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Short Form of Nepean Dyspepsia Index (SF-NDI) | Screening, day 30 and day 60
  The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study). Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
  The total score gives an overall measure of the impact of dyspepsia on the individual, with higher scores indicating more severe symptoms or greater impairment in quality of life due to dyspepsia.
COPE Questionnaire | Screening, day 30 and day 60
  Problem-Focused Coping: A high score indicates coping strategies that are aimed at changing the stressful situation. High scores are indicative of psychological strength, grit, a practical approach to problem solving and is predictive of positive outcomes.
  Emotion-Focused Coping: A high score indicates coping strategies that are aiming to regulate emotions associated with the stressful situation. High or low scores are not uniformly associated with psychological health or ill health, but can be used to inform a wider formulation of the respondent's coping styles.
  Avoidant Coping: A high score indicates physical or cognitive efforts to disengage from the stressor. Low scores are typically indicative of adaptive coping.
Gastrointestinal Symptom Rating Scale (GSRS) | Screening, day 30 and day 60
  The GSRS contains 15 items. All individual items are scored on a 7-point Likert scale (1 = not at all to 7 = extremely) and are subsequently clustered into five domains (abdominal pain, reflux, indigestion, diarrhea, and constipation); higher scores indicate more severe symptoms.
Time required to relief pain for acid reflux flare/heartburn symptoms | Screening, day 30 and day 60
  Participants should consume the investigational product during an acid reflux flare-up or heartburn and record the time taken to achieve relief.
  The time will be recorded.
STAI (State-Trait Anxiety Inventory) | Screening and day 60
  STAI: State-Trait-Anxiety-Inventory-Score This test consists of 20 items and assesses the current state of anxiety in relation to the current situation in which the patient is to the current situation in which the patient finds herself (State Anxiety) and the general anxiety state existing state of anxiety, which represents a part of her personality (Trait Anxiety).
  The sum score has a range from 20-80. Its interpretation with respective score are discussed below:
  mild anxiety (20 to 39); moderate anxiety (40 to 59); intense anxiety (60 to 80).
Profile of Mood State (POMS) questionnaire | Screening and day 60
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 40 item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "Extremely". Higher score indicates worse mood. Total POMS score categories and stress inference:
  0-40 = A little; 81-120= Quite a lot; 41-80= Moderately; 121-160= Extremely.
Change in serum cortisol levels | Screening, day 15 and day 60
  The cortisol secretion will be evaluated by measuring morning serum cortisol levels
Changes in 7 point Likert scale scores | Screening, day 15, 30 and day 60
  The score of patients on the degree of remission of gastroesophageal reflux disease symptoms (acid reflux and heartburn) 1 - No discomfort at all, 2- Minor discomfort, 3- Mild discomfort, 4- Moderate discomfort, 5- Moderately severe discomfort, 6- Severe discomfort, 7- Very severe discomfort

SECONDARY OUTCOMES:
Safety of participant Assessed using adverse events | Screening, baseline, day 15, day 30, day 60
  It is measure in terms of No. of events parameters.
Safety of participant Assessed using treatment compliance and tolerability of investigational product | Screening, baseline, day 15, day 30, day 60
  It is measure in terms of percentage
Systolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Diastolic blood pressure difference from reference measurement (mmHg) | Screening, baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Pulse rate difference from reference measurement (beats per minute) | Screening, baseline, day 15, day 30, day 60
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Complete blood count | Screening and day 60
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)] Red blood cell count [Millions per microliter (million/uL)]
Serum Glutamic Pyruvic Transaminase (SGPT) | Screening and day 60
  Blood level of SGPT was measured. (U/L)
Serum glutamic-oxaloacetic transaminase (SGOT) | Screening and day 60
  Blood level of SGOT was measured. (U/L)
Creatinine difference from reference measurement (mg/dl) | Screening and day 60
  Blood levels of Creatinine was measured. (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramshyam Agarwal, MBBS, DNB, Principal Investigator — Lokmanya Medical Research Centre and Hospital

IPD SHARING:
Plan to Share IPD: No